CLINICAL TRIAL: NCT03275428
Title: Efficacy and Safety of Transnasal Humidified Rapid-insufflation Ventilator Exchange (THRIVE) and Non-intubated Thoracic Surgery (NITS)
Brief Title: THRIVE and Non-intubated Thoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-07-002B
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Thoracic Surgery; Oxygenation
Keywords: THRIVE; Non-intubated thoracic surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- THRIVE group: Patients receiving non-intubated thoracic surgery for lung nodule resections using intravenous sedation and transnasal humidified rapid-insufflation ventilator exchange
  Interventions: Device: transnasal humidified rapid-insufflation ventilator exchange
- Double lumen group: Patients receiving non-intubated thoracic surgery for lung nodule resections using general anesthesia and double lumen endobronchial tube

INTERVENTIONS:
Device: transnasal humidified rapid-insufflation ventilator exchange — high flow nasal cannula with humidified oxygen
  Groups: THRIVE group

SUMMARY:
Video assisted thoracic surgery utilizes small instruments to perform complicated thoracic surgeries. This minimally invasive technique leaves small wounds thus facilitate recovery. Traditionally, thoracic surgery required general anesthesia with double lumen endobronchial tube to facilitate one-lung ventilation. However, as anesthesia techniques improve, video assisted thoracic surgery can be achieved with minimal sedation and without intubation. Thoracic surgeries involve excision of lung tissue thus impair post-operative lung function, putting patients at high risk of cardiopulmonary complications. Non-intubate thoracic surgeries can avoid this complication by avoiding general anesthesia and intubation.

Transnasal humidified rapid-insufflation ventilator exchange offers 30-50 L/min oxygen via nasal cannula, thus provide safe and comfortable way of oxygen supplementation. It is useful in intravenous sedated patients since they are prone to hypoxia from respiratory suppression and upper airway obstruction.

This study is a matched case-control study to compare the efficacy and safety of Transnasal humidified rapid-insufflation ventilator exchange in non-intubated thoracic surgery versus double lumen endobronchial tube intubated general anesthesia.

DETAILED DESCRIPTION:
Lung cancer has been a leading cause of death for years. There are more than 10,000 new cases in Taiwan. Delayed discovery of the disease is a reason for high mortality rate. Most cases are discovered after second stage. Early discovery of the disease rely on low dose CT scans. Early stage lung cancer patients are candidates for minimally invasive surgeries. Traditionally thoracomies and video-assisted thoracic surgeries require general anesthesia with double lumen endobronchial tubes. The technique of double lumen intubation and one lung ventilation causes respiratory complications and damage to the trachea, larynx and vocal cords. With the development of single port thoracotomies, anesthesia can be minimized as well. Patients receive an epidural, intercostal or paravertebral nerve block to decrease pain. Minimal anesthetic agents may be given to decrease anxiety or to induce light sedation. Patients does not need to be intubated and can maintain respiratory function and can recover quickly.

Not only can video-assisted thoracic surgery be used in lung tumor treatment, it can also be used to threat esophageal and mediastinal lesions, pneumothorax or as a diagnostic tool. Video-assisted thoracic surgery was shown to decrease acute phase inflammatory reactions, decrease immunosuppression and can be beneficial for tumor treatment.

The intravenous sedation medications used in non-intubate thoracic surgery decrease pain and anxiety. However, many will develop respiratory depression and upper airway obstruction. Also, spontaneous pneumothorax during surgery causes one lung ventilation. Traditional oxygen supply cannot meet the demand of non-intubated thoracic surgery. Transnasal humidified rapid-insufflation ventilator exchange offers 30-70 L/min oxygen via nasal cannula. Its humidified oxygen can decrease discomfort from cold dry gas. It also provides positive pressure to the airway thus decrease airway obstruction.

Our hypothesis is that non-intubated thoracic surgery with transnasal humidified rapid-insufflation ventilator exchange can maintain optimal surgical condition such as maintain arterial oxygen pressure, decrease acute phase reactions, tumor suppression and accelerate recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Lung nodules requiring surgical resection
* Resectable by video-assisted thoracic surgery

Exclusion Criteria:

* ASA class IV or V
* Room air oxygen saturation by pulse oximeter < 90%
* Emergent surgery
* Use of inotropics or vasoconstrictors
* History of nasal surgery or cranial surgery
* Abnormal coagulation profile
* History of spinal surgery or trauma

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung nodules requiring surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-09-11 (Estimated); Primary Completion 2018-09-10 (Estimated); Study Completion 2018-09-10 (Estimated)

PRIMARY OUTCOMES:
Arterial oxygen pressure | From induction of anesthesia to surgical procedure to end of recovery room observation, duration of six hours.
  Capability of maintaining arterial oxygen pressure > 100 mmHg from arterial blood gas analysis before anesthetic induction, during surgery and in recovery room.
Arterial carbon dioxide pressure | From induction of anesthesia to surgical procedure to end of recovery room observation, duration of six hours.
  Capability of maintaining arterial carbon dioxide pressure < 50 mmHg from arterial blood gas analysis before anesthetic induction, during surgery and in recovery room.
Duration of stay | From admission to ward to discharge from ward, duration of 5 days to two weeks.
  Duration of stay as in days of admission in the hospital

SECONDARY OUTCOMES:
Acute phase reaction | From induction of anesthesia to surgical procedure to fifth post-operative day, duration of six days.
  Measure of C-reactive protein from blood sample analysis before anesthetic induction, after tumor resection during surgery, on post-operative day 1, 3 and 5.
Interleukins | From induction of anesthesia to surgical procedure to fifth post-operative day, duration of six days.
  Measure of interleukins from blood sample analysis before anesthetic induction, after tumor resection during surgery, on post-operative day 1, 3 and 5.
TNF | From induction of anesthesia to surgical procedure to fifth post-operative day, duration of six days.
  Measure of interleukins from blood sample analysis before anesthetic induction, after tumor resection during surgery,
Immune cell count | From induction of anesthesia to surgical procedure to fifth post-operative day, duration of six days.
  Measure of Immune cell count from blood sample analysis before anesthetic induction, after tumor resection during surgery,

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Kun Ting, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Department of Anesthesiology, Taipei Veterans General Hospital, Taipei, Taiwan